CLINICAL TRIAL: NCT05610423
Title: Covid-19 Vaccine Associated Myocarditis and Pericarditis in Norway
Status: Enrolling by invitation | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Norwegian Medicines Agency (Other Government)
Responsible Party: Principal Investigator, Nina Eide Hasselberg, Consultant cardiologist, Oslo University Hospital
Other Study IDs: 434476
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Myocarditis
Keywords: Vaccine side effect; Long term cardiac follow up
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood will be drawn from study participants for routine biochemistry. By separate consent from participants, blood will be stored in a study specific biobank pending analyses, including genetic analyses by whole genome sequencing to search for genetic variants associated with vaccine associated myocarditis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 vaccine associated myocarditis: No intervention
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention. Observational study only

SUMMARY:
This is a national multicenter study in Norway investigating of individuals with Covid-19 vaccine associated myocarditis (VAM) and pericarditis in Norway.

The main objective is to validate the reported possible cases of Covid-19 vaccine associated myo-and pericarditis in Norway as well as investigate for predisposing factors and risk factors for developing these vaccine adverse events.

Furthermore, patients with confirmed Covid-19 VAM, will be invited to participate in a prospective cohort study, investigating for cardiac long-term adverse effects 1 year and 2 years after vaccine-associated myocarditis.

DETAILED DESCRIPTION:
Myocarditis and pericarditis following vaccination with Covid-19 vaccines has been reported as rare but unexpected and potentially severe vaccine adverse events.

In Norway, all vaccines administrated are registered in the national vaccine registry (SYSVAK). All in-hospital diagnoses are reported in a national diagnosis registry (NPR). These complete national high-quality registers allow linking diagnosis of myocarditis and pericarditis to vaccine data (date, product, dose number) on an individual level.

Oslo University Hospital, in collaboration with the Norwegian Institute of Public Health and the Norwegian Medicines Agency, will perform a study consisting of 2 parts:

Part 1 "Validation study":

Eligible patients for inclusion are all individuals with suspected / reported Covid - 19 vaccine associated pericarditis and myocarditis in Norway from 2021 and onwards. Patients will be identified by linking data from the Norwegian Patient registry NPR (ICD-10 diagnostic codes for pericarditis and myocarditis) and the Immunization registry (SYSVAK) (< 90 days since vaccination). The diagnosis of Covid-19 vaccine associated pericarditis and myocarditis will then be confirmed or rejected by medical record search according to international accepted Brighton criteria. The Brighton collaboration criteria provide evidence levels of diagnostic certainty of myocarditis and pericarditis based on cardiac signs and symptoms, cardiac enzymes, ECG findings, imaging studies and histopathology.The criteria is used to distinguish between suspected, probable and confirmed diagnosis of myocarditis and pericarditis. Patients with another more likely reason for confirmed myocarditis or pericarditis by Brighton will not be classified with Covid-19 vaccine associated myocarditis (VAM) or pericarditis, respectively.

Part 2 "Clinical follow-up study" All patients identified in the validation study with confirmed Covid-19 VAM will be invited to participate in the prospective clinical follow-up study (all age groups, both sexes, all geographical areas of Norway). Inclusion wil be by informed consent. Data collection, symptom reporting and cardiac examinations (clinical examination, ECG, 24 hours Holter ECG, echocardiography, cardiac magnetic resonance imaging) will be performed at 1 and 2 years after a diagnosis of Covid -19 VAM. Blood analyses will be performed and a blood sample stored in a biobank in consenting participants. Clinical endpoints will be collected at 1 and 2 years follow-up.

ELIGIBILITY:
Part 1 Individuals identified with possible Covid-19 vaccine associated myocarditis and pericarditis, by linkage of diagnosis of myocarditis and pericarditis (from Norwegian Patient Registry, NPR) and vaccination data (Immunization registry, SYSVAK).

Part 2.

Inclusion Criteria:

* Confirmed myocarditis (definite, probable, possible) by Brighton criteria < 90 days after either Covid-19 vaccine.

Exclusion Criteria:

* Other more likely cause of myocarditis, including Covid-19 infection.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Covid-19 vaccine associated myocarditis and pericarditis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of myocardial scar | 1 year post myocarditis
  Quantification of myocardial scar by cardiac magnetic resonance (CMR).
Reduced myocardial function | 1 year post myocarditis
  Assessment of myocardial function by echocardiography and CMR
Presence of supraventricular arrhythmias | 1 year post myocarditis
  Presence, frequency and type supraventricular arrhythmias detected on ECG and 24 hours Holter ECG recording
Presence of ventricular arrhythmias | 1 year post myocarditis
  Presence, frequency and type of ventricular arrhythmias detected on ECG and 24 hours Holter ECG
Persisting cardiac symptoms. | 2 years post myocarditis
  Participant reporting shortness of breath,chest pain, dizziness, syncope, fatigue.
All cause death | 1 year post myocarditis
  Register death by cause

SECONDARY OUTCOMES:
Presence of myocardial scar | 2 years post myocarditis
  Quantification of myocardial scar by cardiac magnetic resonance (CMR).
Reduced myocardial function | 2 years post myocarditis
  Assessment of myocardial function by echocardiography and CMR
Presence of supraventricular arrhythmias | 2 years post myocarditis
  Presence, frequency and type supraventricular arrhythmias detected on ECG and 24
Presence of ventricular arrhythmias | 2 years post myocarditis
  Presence, frequency and type of ventricular arrhythmias detected on ECG and 24 hours
Persisting cardiac symptoms. | 2 years post myocarditis
  Participant reporting shortness of breath,chest pain, dizziness, syncope, fatigue.
All cause death | 2 years post myocarditis
  Register death by cause

CONTACTS AND LOCATIONS:
Overall Officials: Nina E Hasselberg, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No